CLINICAL TRIAL: NCT02574078
Title: A Master Protocol of Phase 1/2 Studies of Nivolumab in Advanced NSCLC Using Nivolumab as Maintenance After Induction Chemotherapy or as First-line Treatment Alone or in Combination With Standard of Care Therapies (CheckMate 370: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 370)
Brief Title: A Study of Nivolumab in Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: CheckMate370
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-370
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Bevacizumab; Pemetrexed; 130-nm albumin-bound paclitaxel; Paclitaxel; Docetaxel; Gemcitabine; Erlotinib Hydrochloride; Crizotinib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group A Nivolumab (Experimental): Opdivo specified dose on specified days
  Interventions: Drug: Nivolumab
- Group A Nivolumab + SOC maintenance therapy (Experimental): Opdivo/Bevacizumab specified dose on specified days
  Opdivo/Pemetrexed specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Bevacizumab; Drug: Pemetrexed
- Group A SOC maintenance therapy (Active Comparator): Bevacizumab specified dose on specified days
  Pemetrexed specified dose on specified days
  Interventions: Drug: Bevacizumab; Drug: Pemetrexed
- Group B Nivolumab (Experimental): Opdivo specified dose on specified days
  Interventions: Drug: Nivolumab
- Group B Best supportive care (Other): Therapy directed against specific symptoms of disease, i.e., palliative radiation or palliative surgery
  Interventions: Other: Best Supportive Care
- Group C Investigator's choice chemotherapy (Active Comparator): Carboplatin/nab-paclitaxel specified dose on specified days
  Carboplatin/paclitaxel specified dose on specified days
  Carboplatin/pemetrexed specified dose on specified days
  Carboplatin/docetaxel specified dose on specified days
  Carboplatin/gemcitabine specified dose on specified days
  Paclitaxel specified dose on specified days
  Docetaxel specified dose on specified days
  Gemcitabine specified dose on specified days
  Pemetrexed specified dose on specified days
  Interventions: Drug: Pemetrexed; Drug: nab-Paclitaxel; Drug: Paclitaxel; Drug: Docetaxel; Drug: Gemcitabine; Drug: Carboplatin
- Group C Nivolumb (Experimental): Opdivo specified dose on specified days
  Interventions: Drug: Nivolumab
- Group D Erlotinib (Active Comparator): Erlotinib specified dose on specified days
  Interventions: Drug: Erlotinib
- Group D Nivolumab + Erlotinib (Experimental): Opdivo/Erlotnib specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Erlotinib
- Group E Nivolumab + Crizotinib (Experimental): Opdivo/Crizotinib specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Crizotinib

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo
  Arms: Group A Nivolumab; Group A Nivolumab + SOC maintenance therapy; Group B Nivolumab; Group C Nivolumb; Group D Nivolumab + Erlotinib; Group E Nivolumab + Crizotinib
Drug: Bevacizumab
  Arms: Group A Nivolumab + SOC maintenance therapy; Group A SOC maintenance therapy
Drug: Pemetrexed
  Arms: Group A Nivolumab + SOC maintenance therapy; Group A SOC maintenance therapy; Group C Investigator's choice chemotherapy
Other: Best Supportive Care — Palliative radiation, palliative surgery and/or other best supportive care treatments
  Arms: Group B Best supportive care
Drug: nab-Paclitaxel
  Arms: Group C Investigator's choice chemotherapy
Drug: Paclitaxel
  Arms: Group C Investigator's choice chemotherapy
Drug: Docetaxel
  Arms: Group C Investigator's choice chemotherapy
Drug: Gemcitabine
  Arms: Group C Investigator's choice chemotherapy
Drug: Erlotinib
  Arms: Group D Erlotinib; Group D Nivolumab + Erlotinib
Drug: Crizotinib
  Arms: Group E Nivolumab + Crizotinib
Drug: Carboplatin
  Arms: Group C Investigator's choice chemotherapy

SUMMARY:
The purpose of this study is to determine whether nivolumab monotherapy or in combination with Standard of care (SOC) therapies will provide clinical benefit (i.e., PFS, OS, and DOR) without unacceptable toxicity in advanced Non-Small Cell Lung Cancer patients.

DETAILED DESCRIPTION:
Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK)

**Please note that the study is no longer enrolling patients for Groups A, B, C, and E.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed locally advanced or stage IV NSCLC
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0-2
* Tumor tissue sections must be available for biomarker evaluation

Exclusion Criteria:

* Untreated or active/progressing Central Nervous system (CNS) metastases
* Active, known or suspected autoimmune disease
* Known history of testing positive for HIV or AIDS
* Active or chronic infection of hepatitis B virus or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (132):
- United States (132):
  - Alabama Oncology, Birmingham, Alabama
  - Southern Cancer Center Pc, Mobile, Alabama
  - Arizona Oncology Assoc, Pc-Hal, Glendale, Arizona
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncol Assoc Dba (Hem Onc Physicians&Extenders) Hope, Tucson, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - St. Joseph Heritage Medical Group, Fullerton, California
  - Scripps Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology Clinic, Los Angeles, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Med Oncology, Santa Maria, California
  - Local Institution, Solvang, California
  - St. Mary's Hospital Regional Cancer Center, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Eastern Ct Hem Onc Assoc, Norwich, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Va Ct Healthcare System, West Haven, Connecticut
  - Florida Cancer Specialists S., Fort Myers, Florida
  - University of Florida at Shands, Gainesville, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Baptist Health Medical Group Oncology, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - Florida Cancer Affiliates, Trinity, Florida
  - University Cancer Blood Ctr, Athens, Georgia
  - Cancer Treatment Centers Of America, Newnan, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Ft. Wayne Med Onco-Hema Inc, Fort Wayne, Indiana
  - Cotton-O-Neil Clinical Research Center, Topeka, Kansas
  - West KY Hematology Oncology Group PSC, Paducah, Kentucky
  - Christus St. Francis Cabrini Cancer Center, Alexandria, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University Of Maryland, Baltimore, Maryland
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Center For Cancer And Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - Cancer & Hematology Centers Of Western Michigan, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Forrest General Cancer Center, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Pllc, Jackson, Mississippi
  - St. Louis Cancer Care, Llp, Bridgeton, Missouri
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hunterdon Medical Center, Flemington, New Jersey
  - Summit Medical Group, Morristown, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - Morristown Medical Center, Summit, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - New York Oncology Hematology, Pc, Albany, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Broome Oncology, Johnson City, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Columbia University Medical Center (Cumc), New York, New York
  - Hematology-Oncology Associates Of Rockland, Nyack, New York
  - White Plains Hospital, White Plains, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - Randolph Cancer Center, Greensboro, North Carolina
  - First Health Of The Carolinas, Pinehurst, North Carolina
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Cancer Care Center, Bismarck, North Dakota
  - Sanford Health, Fargo, North Dakota
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mid Ohio Oncology Hematology, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC-Clinical Research, Tulsa, Oklahoma
  - Oncology Associates Of Oregon, Pc, Eugene, Oregon
  - Hematology Oncology Associates, Medford, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's University Hospital Bethlehem, Bethlehem, Pennsylvania
  - Erie Regional Cancer Center, Erie, Pennsylvania
  - Abington Hematology Oncology Associates, Inc, Horsham, Pennsylvania
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Sanford Research, Sioux Falls, South Dakota
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - The Jones Clinic, PC, Germantown, Tennessee
  - West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC - SCRI - PPDS, Nashville, Tennessee
  - Texas Oncology-Abilene, Abilene, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology-Arlington North, Arlington, Texas
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Texas Oncology, Bedford, Texas
  - Texas Oncology/Methodist Charlton Cancer Ctr, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology, Denton, Texas
  - Texas Oncology, El Paso, Texas
  - Texas Oncology, Flower Mound, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Oncology, Fort Worth, Texas
  - The Center For Cancer And Blood Disorders, Fort Worth, Texas
  - Texas Oncology, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Cancer Center Of Mesquite, Mesquite, Texas
  - Texas Oncology, Pa, Midland, Texas
  - Texas Oncology, New Braunfels, Texas
  - Texas Oncology, Paris, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology Plano West Cancer Center, Plano, Texas
  - Cancer Centers of South Texas, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology Cancer Center - Sugar Land, Sugar Land, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology Cancer Care And Research Center, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Texas Oncology, Weslaco, Texas
  - Texas Oncology-Wichita Falls, Wichita Falls, Texas
  - Oncology & Hematology Associates Of Southwest Virginia, Inc., Blacksburg, Virginia
  - Virginia Cancer Specialists, Pc, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Shenandoah Oncology, Winchester, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - Northwest Cancer Specialists, Pc, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 341 participants were grouped as such:
  Groups A-D: 328 participants randomized, 314 treated and 14 not treated. Reasons not treated: Group A - 1 no longer met criteria; Group B - 3 withdrew consent, 2 no longer met criteria, 2 other; Group C - 1 no longer met criteria; Group D - 2 withdrew consent, 1 poor/non-compliance, 2 other.
  Group E: 13 participants treated.
Groups:
- Group A, Cohort A, Nivo; Group A, Cohort B, Nivo; Group B, Nivo; Group C, Nivo: Nivolumab 240 mg every 2 weeks.
- Group A, Cohort A, Beva + Nivo: Bevacizumab 15 mg/kg + nivolumab 5 mg/kg every 3 weeks.
- Group A, Cohort A, Beva: Bevacizumab 15 mg/kg every 3 weeks.
- Group A, Cohort B, Peme + Nivo: Pemetrexed 500 mg/m^2 every 3 weeks + nivolumab 5 mg/kg every 3 weeks.
- Group A, Cohort B, Peme: Pemetrexed 500 mg/m^2 every 3 weeks.
- Group B, BSC: Best Supportive Care (BSC)
- Group C, ICC: Investigator's Choice of Chemotherapy
- Group D, Nivo + Erlo: Nivolumab 240 mg every 2 weeks + erlotinib 150 mg once a day (QD).
- Group D, Erlo: Erlotinib 150 mg QD.
- Group E: Nivolumab 240 mg every 2 weeks + crizotinib 250 mg two times a day (BID).
Period: Pre-Treatment Period
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo | Group E
Started (Started = Randomized (entering treatment)) | 13 | 6 | 9 | 35 | 34 | 35 | 18 | 17 | 26 | 26 | 53 | 56 | 13
Completed (Finished = Treated) | 13 | 6 | 9 | 35 | 34 | 34 | 14 | 14 | 25 | 26 | 49 | 55 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 1 | 0 | 4 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Poor/non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Treatment Period
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo | Group E
Started (Started = Treated) | 13 | 6 | 9 | 35 | 34 | 34 | 14 | 14 | 25 | 26 | 49 | 55 | 13
Completed | 3 | 0 | 0 | 7 | 3 | 1 | 2 | 2 | 1 | 9 | 4 | 8 | 0
Not Completed | 10 | 6 | 9 | 28 | 31 | 33 | 12 | 12 | 24 | 17 | 45 | 47 | 13
Not completed — Disease progression | 6 | 4 | 7 | 18 | 16 | 26 | 5 | 9 | 8 | 5 | 20 | 29 | 2
Not completed — Study drug toxicity | 1 | 1 | 0 | 5 | 3 | 1 | 2 | 0 | 2 | 1 | 16 | 2 | 4
Not completed — Death | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 7 | 1 | 0 | 2 | 1
Not completed — Adverse event unrelated to drug | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 0 | 1 | 2 | 4 | 1 | 0
Not completed — Administrative reason by Sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Other reasons | 1 | 0 | 1 | 3 | 3 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 1
Not completed — Participant request to stop drug | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 3 | 2 | 2 | 4 | 1
Not completed — Participant withdrew consent | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 4 | 1
Not completed — Participant no longer meets criteria | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo | Group E | Total
Number analyzed (Participants) | 13 | 6 | 9 | 35 | 34 | 35 | 18 | 17 | 26 | 26 | 53 | 56 | 13 | 341
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 8 | 2 | 1 | 15 | 14 | 15 | 5 | 4 | 3 | 4 | 21 | 20 | 7 | 119
  >= 65 and < 75 years old | 4 | 2 | 3 | 15 | 13 | 15 | 10 | 9 | 13 | 11 | 21 | 24 | 1 | 141
  >= 75 years old | 1 | 2 | 5 | 5 | 7 | 5 | 3 | 4 | 10 | 11 | 11 | 12 | 5 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 21 | 13 | 21 | 11 | 9 | 12 | 14 | 33 | 31 | 6 | 185
  Male | 7 | 2 | 5 | 14 | 21 | 14 | 7 | 8 | 14 | 12 | 20 | 25 | 7 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 1 | 3 | 5 | 0 | 17
  Not Hispanic or Latino | 13 | 6 | 8 | 34 | 31 | 32 | 17 | 16 | 26 | 23 | 50 | 51 | 13 | 320
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 10 | 1 | 22
  Black or African American | 3 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 3 | 4 | 2 | 2 | 1 | 22
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 9 | 6 | 7 | 31 | 32 | 34 | 16 | 15 | 23 | 21 | 41 | 43 | 10 | 288
  Other | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), Groups A-D Only
Description: Progression-free survival (PFS) is defined as the time from randomization to the date of the first documented tumor progression, as determined by investigators (per RECIST v1.1), or death due to any cause, whichever occurs first.
Time Frame: up to approximately 48 months
Population: All randomized participants in Groups A-D only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo
Number analyzed (Participants) | 13 | 6 | 9 | 35 | 34 | 35 | 18 | 17 | 26 | 26 | 53 | 56
Months | 15.0 [1.4 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 6.7 [4.1 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 6.0 [3.3 to 19.3] | 5.9 [2.6 to 12.9] | 8.1 [4.0 to 12.0] | 5.0 [2.1 to 6.8] | 9.6 [2.1 to 24.2] | 2.3 [1.0 to 4.0] | 2.7 [1.2 to 4.9] | 6.7 [4.4 to 13.1] | 11.0 [9.3 to 17.0] | 11.0 [7.6 to 13.0]
Statistical Analysis 1: Comparison: Group A, Cohort A, Nivo vs Group A, Cohort A, Beva; Test type: Superiority; p = 0.5050, Unstratified log-rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.24 to 2.03]
Statistical Analysis 2: Comparison: Group A, Cohort A, Beva + Nivo vs Group A, Cohort A, Beva; Test type: Superiority; p = 0.6284, Unstratified log-rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.22 to 2.54]
Statistical Analysis 3: Comparison: Group A, Cohort B, Nivo vs Group A, Cohort B, Peme; Test type: Superiority; p = 0.1988, Unstratified log-rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.40 to 1.22]
Statistical Analysis 4: Comparison: Group A, Cohort B, Peme + Nivo vs Group A, Cohort B, Peme; Test type: Superiority; p = 0.2722, Unstratified log-rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.42 to 1.28]
Statistical Analysis 5: Comparison: Group B, Nivo vs Group B, BSC; Test type: Superiority; p = 0.0544, Unstratified log-rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.17 to 1.04]
Statistical Analysis 6: Comparison: Group C, Nivo vs Group C, ICC; Test type: Superiority; p = 0.0442, Unstratified log-rank; Hazard Ratio (HR) = 2.04, 95% CI 2-sided [1.00 to 4.16]
Statistical Analysis 7: Comparison: Group D, Nivo + Erlo vs Group D, Erlo; Test type: Superiority; p = 0.5489, Log Rank; stratified by Disease Status (Recurrent Locally Advanced vs. Metastatic), Performance Status (ECOG 0 vs.1 vs. 2) as entered into the IVRS; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.50 to 1.45]

2. Primary Outcome: Overall Survival (OS), Groups A-C Only
Description: Overall survival (OS) is defined as the time from randomization to the date of death.
Time Frame: up to approximately 60 months
Population: All randomized participants in Groups A-C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC
Number analyzed (Participants) | 13 | 6 | 9 | 35 | 34 | 35 | 18 | 17 | 26 | 26
Months | 20.0 [2.4 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 30.8 [8.8 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 18.1 [3.3 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 28.9 [14.8 to 38.3] | 17.4 [10.7 to 39.7] | 18.4 [6.7 to 30.9] | NA [11.0 to NA] — Median not reached as insufficient progression events among responders | 13.6 [2.0 to 36.8] | 3.9 [1.5 to 12.5] | 15.8 [6.5 to 23.1]
Statistical Analysis 1: Comparison: Group A, Cohort A, Nivo vs Group A, Cohort A, Beva; Test type: Superiority; p = 0.9951, Unstratified log-rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.35 to 2.91]
Statistical Analysis 2: Comparison: Group A, Cohort A, Beva + Nivo vs Group A, Cohort A, Beva; Test type: Superiority; p = 0.8321, Unstratified log-rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.25 to 3.10]
Statistical Analysis 3: Comparison: Group A, Cohort B, Nivo vs Group A, Cohort B, Peme; Test type: Superiority; p = 0.2938, Unstratified log-rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.41 to 1.31]
Statistical Analysis 4: Comparison: Group A, Cohort B, Peme + Nivo vs Group A, Cohort B, Peme; Test type: Superiority; p = 0.4819, Unstratified log-rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.46 to 1.45]
Statistical Analysis 5: Comparison: Group B, Nivo vs Group B, BSC; Test type: Superiority; p = 0.0241, Unstratified log-rank; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.11 to 0.91]
Statistical Analysis 6: Comparison: Group C, Nivo vs Group C, ICC; Test type: Superiority; p = 0.1401, Unstratified log-rank; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.85 to 2.95]

3. Primary Outcome: Percentage of Participants With Treatment-related Adverse Events (AEs) Leading to Both Study Drugs Discontinuation, Group E Only
Description: Percentage of participants who experienced a treatment-related AE during the course of the study that lead to discontinuation of both study drugs.
Time Frame: up to approximately 60 months
Population: All treated participants in Group E only
Measure: Number; unit: Percentage of participants
Arm/Group | Group E
Number analyzed (Participants) | 13
Percentage of participants | 38.5

4. Secondary Outcome: Duration of Response (DOR), Groups A-D Only
Description: Duration of response (DOR) is defined as the time from first confirmed response (complete response (CR) or partial response (PR)) to the date of the initial objectively documented tumor progression as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first.
  Median computed using Kaplan-Meier method.
Time Frame: up to approximately 48 months
Population: All responders (participants with objective response of CR or PR) in Groups A-D only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo
Number analyzed (Participants) | 3 | 1 | 1 | 10 | 7 | 1 | 3 | 1 | 5 | 4 | 33 | 35
months | 12.780 [4.140 to 20.435] | NA [NA to NA] — Median not reached as insufficient progression events among responders | 17.084 [NA to NA] — only 1 participant | 12.912 [1.873 to 31.113] | 8.542 [2.464 to 9.265] | 14.982 [NA to NA] — only 1 participant | NA [11.072 to NA] — Median not reached as insufficient progression events among responders | NA [NA to NA] — Median not reached as insufficient progression events among responders | 3.877 [2.103 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 2.940 [1.577 to 4.304] | 8.805 [5.520 to 13.437] | 10.152 [5.552 to 17.314]

5. Secondary Outcome: Objective Response Rate (ORR), Groups A-E
Description: Objective response rate (ORR) is defined as the number and percentage of participants with a best overall response (BOR) of confirmed complete response (CR) or partial response (PR). Best overall response (BOR) is defined as the best response designation, recorded between the date of first dose and the date of the initial objectively documented tumor progression per RECIST v1.1 or the date of subsequent therapy, whichever occurs first.
  Confidence interval based on the Clopper and Pearson method.
Time Frame: up to approximately 48 months
Population: All randomized (Groups A-D) and treated (Group E) participants with at least one lesion at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A, Cohort A, Nivo | Group A, Cohort A, Beva + Nivo | Group A, Cohort A, Beva | Group A, Cohort B, Nivo | Group A, Cohort B, Peme + Nivo | Group A, Cohort B, Peme | Group B, Nivo | Group B, BSC | Group C, Nivo | Group C, ICC | Group D, Nivo + Erlo | Group D, Erlo | Group E
Number analyzed (Participants) | 13 | 6 | 8 | 34 | 33 | 32 | 16 | 17 | 24 | 26 | 51 | 56 | 13
Percentage of participants | 23.1 [5.0 to 53.8] | 16.7 [0.4 to 64.1] | 12.5 [0.3 to 52.7] | 29.4 [15.1 to 47.5] | 21.2 [9.0 to 38.9] | 3.1 [0.1 to 16.2] | 18.8 [4.0 to 45.6] | 5.9 [0.1 to 28.7] | 20.8 [7.1 to 42.2] | 15.4 [4.4 to 34.9] | 64.7 [50.1 to 77.6] | 62.5 [48.5 to 75.1] | 23.1 [5.0 to 53.8]

6. Secondary Outcome: Overall Survival (OS), Group D Only
Description: Overall survival (OS) is defined as the time from randomization to the date of death.
Time Frame: up to approximately 60 months
Population: All randomized participants in Group D only
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group D, Nivo + Erlo | Group D, Erlo
Number analyzed (Participants) | 53 | 56
months | NA [23.1 to NA] — Median not reached as insufficient progression events among responders | 34.8 [22.5 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold
Statistical Analysis 1: Comparison: Group D, Nivo + Erlo vs Group D, Erlo; Test type: Superiority; p = 0.2862, Log Rank; [statistical method as in outcome 1, analysis 7]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.40 to 1.31]

7. Secondary Outcome: Progression-Free Survival (PFS), Group E Only
Description: as for outcome 1
Time Frame: up to approximately 48 months
Population: All treated participants in Group E only
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group E
Number analyzed (Participants) | 13
months | 9.63 [0.95 to 20.11]

ADVERSE EVENTS:
Time Frame: Treated population: From first dose to 100 days post last dose (approximately 60 months)
Groups:
- SUB-STUDY A, COHORT A: NIVOLUMAB 240 MG; SUB-STUDY A, COHORT B: NIVOLUMAB 240 MG; SUB-STUDY B: NIVOLUMAB 240 MG; SUB-STUDY C: NIVOLUMAB 240 MG: Nivolumab 240 mg every 2 weeks.
- SUB-STUDY A: BEVACIZUMAB + NIVOLUMAB 5 MG/KG: Bevacizumab 15 mg/kg + nivolumab 5 mg/kg every 3 weeks.
- SUB-STUDY A: BEVACIZUMAB: Bevacizumab 15 mg/kg every 3 weeks.
- SUB-STUDY A: PEMETREXED + NIVOLUMAB 5 MG/KG: Pemetrexed 500 mg/m^2 every 3 weeks + nivolumab 5 mg/kg every 3 weeks.
- SUB-STUDY A: PEMETREXED: Pemetrexed 500 mg/m^2 every 3 weeks.
- SUB-STUDY B: BEST SUPPORTIVE CARE: Best Supportive Care (BSC)
- SUB-STUDY C: INVESTIGATOR'S CHOICE OF CHEMOTHERAPY: Investigator's Choice of Chemotherapy (ICC)
- SUB-STUDY D: NIVOLUMAB 240 MG + ERLOTINIB: Nivolumab 240 mg every 2 weeks + erlotinib 150 mg once a day (QD).
- SUB-STUDY D: ERLOTINIB: Erlotinib 150 mg QD.
- SUB-STUDY E: SINGLE ARM: NIVOLUMAB 240 MG + CRIZOTINIB: Nivolumab 240 mg every 2 weeks + crizotinib 250 mg two times a day (BID).
Arm/Group | SUB-STUDY A, COHORT A: NIVOLUMAB 240 MG | SUB-STUDY A: BEVACIZUMAB + NIVOLUMAB 5 MG/KG | SUB-STUDY A: BEVACIZUMAB | SUB-STUDY A, COHORT B: NIVOLUMAB 240 MG | SUB-STUDY A: PEMETREXED + NIVOLUMAB 5 MG/KG | SUB-STUDY A: PEMETREXED | SUB-STUDY B: NIVOLUMAB 240 MG | SUB-STUDY B: BEST SUPPORTIVE CARE | SUB-STUDY C: NIVOLUMAB 240 MG | SUB-STUDY C: INVESTIGATOR'S CHOICE OF CHEMOTHERAPY | SUB-STUDY D: NIVOLUMAB 240 MG + ERLOTINIB | SUB-STUDY D: ERLOTINIB | SUB-STUDY E: SINGLE ARM: NIVOLUMAB 240 MG + CRIZOTINIB
All-Cause Mortality (participants affected / at risk) | 8/13 | 4/6 | 6/9 | 24/35 | 23/34 | 24/34 | 5/14 | 9/14 | 23/25 | 18/26 | 20/49 | 25/55 | 7/13
Serious Adverse Events (participants affected / at risk) | 6/13 | 1/6 | 5/9 | 15/35 | 16/34 | 14/34 | 5/14 | 7/14 | 23/25 | 7/26 | 25/49 | 17/55 | 8/13
Other Adverse Events (participants affected / at risk) | 12/13 | 6/6 | 9/9 | 35/35 | 32/34 | 33/34 | 13/14 | 13/14 | 22/25 | 25/26 | 49/49 | 55/55 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUB-STUDY A, COHORT A: NIVOLUMAB 240 MG (N=13) | SUB-STUDY A: BEVACIZUMAB + NIVOLUMAB 5 MG/KG (N=6) | SUB-STUDY A: BEVACIZUMAB (N=9) | SUB-STUDY A, COHORT B: NIVOLUMAB 240 MG (N=35) | SUB-STUDY A: PEMETREXED + NIVOLUMAB 5 MG/KG (N=34) | SUB-STUDY A: PEMETREXED (N=34) | SUB-STUDY B: NIVOLUMAB 240 MG (N=14) | SUB-STUDY B: BEST SUPPORTIVE CARE (N=14) | SUB-STUDY C: NIVOLUMAB 240 MG (N=25) | SUB-STUDY C: INVESTIGATOR'S CHOICE OF CHEMOTHERAPY (N=26) | SUB-STUDY D: NIVOLUMAB 240 MG + ERLOTINIB (N=49) | SUB-STUDY D: ERLOTINIB (N=55) | SUB-STUDY E: SINGLE ARM: NIVOLUMAB 240 MG + CRIZOTINIB (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cyclosporidium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraspinal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 3 | 2 | 0 | 1 | 2 | 1 | 3 | 3 | 2 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 4 | 4 | 3 | 0 | 4 | 8 | 1 | 3 | 5 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUB-STUDY A, COHORT A: NIVOLUMAB 240 MG (N=13) | SUB-STUDY A: BEVACIZUMAB + NIVOLUMAB 5 MG/KG (N=6) | SUB-STUDY A: BEVACIZUMAB (N=9) | SUB-STUDY A, COHORT B: NIVOLUMAB 240 MG (N=35) | SUB-STUDY A: PEMETREXED + NIVOLUMAB 5 MG/KG (N=34) | SUB-STUDY A: PEMETREXED (N=34) | SUB-STUDY B: NIVOLUMAB 240 MG (N=14) | SUB-STUDY B: BEST SUPPORTIVE CARE (N=14) | SUB-STUDY C: NIVOLUMAB 240 MG (N=25) | SUB-STUDY C: INVESTIGATOR'S CHOICE OF CHEMOTHERAPY (N=26) | SUB-STUDY D: NIVOLUMAB 240 MG + ERLOTINIB (N=49) | SUB-STUDY D: ERLOTINIB (N=55) | SUB-STUDY E: SINGLE ARM: NIVOLUMAB 240 MG + CRIZOTINIB (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 4 | 11 | 8 | 0 | 2 | 3 | 5 | 16 | 10 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 8 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 5 | 3 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 6 | 1 | 1 | 3 | 0 | 2 | 0 | 5 | 4 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 7 | 7 | 0
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 3 | 1 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 3 | 2 | 2 | 0 | 6 | 1 | 6 | 6 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 6 | 7 | 3 | 4 | 1 | 5 | 5 | 8 | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 5 | 13 | 9 | 3 | 5 | 1 | 7 | 9 | 33 | 36 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 5 | 1 | 0 | 0 | 1 | 2 | 5 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 4 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 3 | 0 | 4 | 4 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 2 | 7 | 8 | 9 | 2 | 0 | 8 | 10 | 24 | 21 | 6
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 10 | 9 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 3 | 4 | 1 | 2 | 4 | 4 | 10 | 10 | 4
Asthenia (General disorders) | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 4 | 4 | 1
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0
Cyst (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 1 | 16 | 13 | 11 | 5 | 2 | 8 | 7 | 25 | 23 | 8
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 2 | 3 | 1 | 1 | 0 | 3 | 0 | 3 | 3 | 0
Oedema peripheral (General disorders) | 1 | 2 | 2 | 4 | 14 | 8 | 0 | 1 | 5 | 5 | 14 | 6 | 5
Pain (General disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 5 | 4 | 6 | 3 | 2 | 3 | 2 | 7 | 1 | 4
Swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 1 | 3 | 3 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 4 | 6 | 2 | 1 | 3 | 1 | 1 | 3 | 7 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 3 | 3 | 3 | 3 | 2 | 1 | 1 | 6 | 2 | 2
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 4 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 4 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 5 | 2 | 2 | 1 | 0 | 1 | 0 | 7 | 6 | 7
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0 | 2 | 2 | 2 | 2 | 0 | 2 | 1 | 6 | 6 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2 | 4 | 4 | 2 | 1 | 2 | 0 | 5 | 2 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Protein total decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 2 | 1 | 1 | 6 | 1 | 1 | 2 | 3 | 4 | 4 | 8 | 5 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 3 | 6 | 11 | 3 | 3 | 2 | 6 | 7 | 15 | 21 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 7 | 10 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0 | 1 | 2 | 2 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 4 | 6 | 3 | 0 | 2 | 2 | 8 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 6 | 4 | 3 | 2 | 3 | 3 | 8 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 1 | 4 | 1 | 1 | 2 | 2 | 3 | 5 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1 | 3 | 2 | 2 | 0 | 1 | 4 | 3 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin C deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 8 | 2 | 0 | 2 | 1 | 1 | 2 | 11 | 5 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 4 | 3 | 5 | 1 | 3 | 5 | 2 | 7 | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 5 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 3 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3 | 0 | 2 | 1 | 1 | 1 | 0 | 5 | 4 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 4 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 2 | 6 | 2 | 0 | 2 | 0 | 2 | 7 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2 | 5 | 0 | 3 | 0 | 1 | 1 | 11 | 4 | 1
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 5 | 8 | 1
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 8 | 4 | 4 | 3 | 1 | 0 | 1 | 8 | 5 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 5 | 2 | 5 | 4 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 5 | 2 | 2 | 2 | 0 | 2 | 0 | 6 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 5 | 2 | 3 | 0 | 1 | 3 | 1 | 9 | 5 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Bladder diverticulum (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2 | 7 | 7 | 7 | 3 | 2 | 4 | 2 | 11 | 14 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 10 | 5 | 6 | 1 | 2 | 5 | 2 | 9 | 10 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 4 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 7 | 10 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 23 | 29 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 11 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 5 | 1 | 2 | 0 | 0 | 0 | 14 | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6 | 2 | 0 | 1 | 0 | 1 | 1 | 9 | 11 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 4 | 2 | 2 | 0 | 2 | 0 | 7 | 10 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 3 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 4 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 2 | 5 | 2 | 1
Jugular vein distension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT02574078/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT02574078/SAP_001.pdf